CLINICAL TRIAL: NCT06279351
Title: Thalidomide Enhances Clinical Efficacy of Cetuximab Combined With Standard Chemotherapy for Left Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director of oncology department, Clinical Professor, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thalicolorectal
Record Dates: First submitted 2023-12-17; First posted 2024-02-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Thalidomide Enhances Clinical Efficacy of Cetuximab Combined With Standard Chemotherapy for Left Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Thalidomide+cetuximab+FOLFOX/FOLFIRI
  Interventions: Drug: Thalidomide+cetuximab+FOLFOX/FOLFIRI
- control group (No Intervention): cetuximab+FOLFOX/FOLFIRI

INTERVENTIONS:
Drug: Thalidomide+cetuximab+FOLFOX/FOLFIRI — Thalidomide+cetuximab+FOLFOX/FOLFIRI
  Arms: Test group

SUMMARY:
1. To verify that thalidomide can increase the efficacy of cetuximab plus chemotherapy in the treatment of stage IV RAS and BRAF wild-type unresectable left colorectal cancer, which has important clinical significance and provides a basis for subsequent large-scale research and clinical application.
2. To evaluate the changes of cytokines and verify the effect of some cytokines on the efficacy of cetuximab +FOLFIRI, so as to provide a scientific basis for the subsequent precise therapy using cytokines antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RAS and BRAF wild-type IV unresectable left colorectal cancer confirmed by pathology and tissue/cytology and genetic testing;
2. Physical state is good: PS 0-2;
3. Expected survival of more than 3 months;
4. Aged 18-75 years old;
5. Have not received systematic chemotherapy before;
6. Did not receive cetuximab treatment;
7. Liver, kidney and bone marrow functions are basically normal;
8. The clearance period of chemotherapy and molecular targeted therapy is more than 4 weeks;
9. Voluntary participation in the group, good compliance, can cooperate with the experiment observation, and sign the written informed consent.

Exclusion Criteria:

1. Patients with severe dysfunction of vital organs (heart, liver, kidney);
2. Patients with other malignant tumors;
3. Patients who are pregnant or breastfeeding (women of childbearing age need to check pregnancy test);
4. In the active phase of acute or chronic infectious diseases;
5. People with a clear history of drug allergy or allergic constitution;
6. Patients participating in other clinical trials;
7. Other conditions in which the patient was considered inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ETS | 8 weeks
  Early tumor shrinkage

SECONDARY OUTCOMES:
ORR | 8 weeks
DCR | 8 weeks
PFS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: rui kong, doctor, Principal Investigator — Chongqing Medical University
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No